CLINICAL TRIAL: NCT01063335
Title: Imaging Cannabinoid CB1 Receptors in Schizophrenia
Status: Terminated | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100058; 10-M-0058
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2012-09-20

CONDITIONS: Schizophrenia
Keywords: CB1 Receptor; Schizophrenia; Positron Emission Tomography (PET); Healthy Volunteers; HV
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- The CB1 receptor is a protein in the brain that is targeted by the active ingredients in cannabis (marijuana). Brain systems that react to cannabis may be involved in the causes and symptoms of schizophrenia and schizoaffective disorder. For instance, research studies have shown that the number of CB1 receptors may be different in people with schizophrenia, and there may be differences in the receptors themselves. Researchers are interested in using positron emission tomography (PET) to study CB1 receptors in people with and without schizophrenia, using a chemical tracer that attaches specifically to CB1 receptors.

Objectives:

- To determine whether the CB1 receptor brain protein is different in people with and without schizophrenia.

Eligibility:

- Individuals between 18 and 55 years of age who either have been diagnosed with schizophrenia/schizoaffective disorder or are healthy volunteers.

Design:

* Participants in the study must have previously enrolled in the National Institute of Mental Health protocol A Neurobiological Investigation of Patients with Schizophrenia Spectrum Disorders and Their Siblings (95-M-0150).
* Participants will provide blood samples to test for the gene that contains information on the specific type of CB1 receptor each participant has.
* Participants will have a PET scan and/or a magnetic resonance imaging (MRI) scan.
* The PET scan will last approximately 2 hours. Participants will receive an injection of a small amount of chemical tracer to improve the quality of the images taken during the scan.
* The MRI scan will last approximately 1 hour.

DETAILED DESCRIPTION:
Schizophrenia is a debilitating mental disorder with a complex and multifactorial etiology. The exact pathophysiological mechanisms have remained elusive, but a large body of evidence points toward abnormalities in a number of brain neurotransmitter systems: dopamine, glutamate, and gamma-amino butyric acid (GABA). Pharmacological studies have shown that acute exposure to cannabis is able to induce psychotic symptoms in healthy individuals and exacerbate symptoms in patients with an established psychotic illness. In addition, epidemiological studies have established that cannabis use in early adolescence is associated with an increased risk of developing schizophrenia later in life. Together, this evidence suggests that the neural systems targeted by cannabis may be involved in the pathophysiology of schizophrenia.

The brain endocannabinoid (EC) system is a recently discovered brain neurotransmission system, which involves endogenous cannabinoid agents (ECs) that act upon specific receptors (CB1 and CB2). CB1 receptor is abundant in the human brain and acts as an inhibitory modulator of classical neurotransmitters. ECs and CB1 receptors appear to be involved in the pathophysiology of schizophrenia. EC levels are elevated in the cerebrospinal fluid of patients with schizophrenia, and post-mortem studies have shown increased density of radioligand binding to brain CB1 receptors. To what extent CB1 receptors are involved in the pathophysiology of schizophrenia in the living human brain is currently unknown. The lack of suitable methods to reliably quantify CB1 receptors in the living human brain have to date hindered the progress in this field.

In this protocol, we outline studies aiming at elucidating the role of CB1 receptors in schizophrenia by using positron emission tomography (PET) and the recently developed radiotracer for CB1 receptors, [18F]FMPEP-d(2). The aim of this project is to explore CB1 receptor abnormalities in human patients with schizophrenia. The primary hypothesis is that CB1 receptor density is increased in patients with schizophrenia in comparison with healthy subjects. Insight into the role of CB1 receptor function in schizophrenia may help guide future development of pharmacotherapies.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with Schizophrenia:

1. All subjects must be 18-55 years of age and be able to give written informed consent.
2. All subjects must be healthy based on history and physical examination.
3. Subjects must fulfill DSM-IV criteria (American Psychiatric Association 1987) for schizophrenia, schizophreniform disorder, or schizo-affective disorder.
4. About half of the patients with schizophrenia will be carriers of the C allele of the rs2023239 SNP and half will not.

Healthy Subjects:

1. All subjects must be18-55 years of age and be able to give written informed consent.
2. This comparison group must be healthy based on history and physical examination.
3. About half of the healthy subjects will currently smoke cigarettes and about half will not. Smoking is defined by daily or near-daily smoking of more than 4 cigarettes/day, and non-smoking is defined by a life-time exposure of less than 100 cigarettes and none in the preceding 2 years.
4. About half of the healthy subjects will be carriers of the C allele of the rs2023239 SNP and half will not.

EXCLUSION CRITERIA:

Patients with Schizophrenia:

1. Any serious medical condition as judged by the Principal Investigator.
2. The patient has a guardian or a Durable Power of Attorney.
3. Past or present diagnosis of primary mood disorders (such as bipolar illness or major depressive disorder). Any present substance abuse. Cannibis use within the last 2 months.
4. Diagnosis of alcohol abuse or alcohol dependence as defined by DSM-IV (American Psychiatric Association 1987) criteria. Recent heavy use of alcohol. That is, subjects must have an alcohol audit score of less than or equal to 9. In addition, subjects must agree not to consume any alcohol in the three days prior to the PET scan.
5. Positive test for HIV.
6. Metallic foreign bodies that would be affected by the MRI scanner magnet, or fear of enclosed spaces likely to make the subject unable to undergo an MRI scan.
7. Head trauma resulting in a period of unconsciousness lasting longer than 1 hour.
8. History of fetal alcohol syndrome or other neurodevelopmental disorder.
9. History of seizures, other than in childhood and related to fever.
10. Recent exposure to radiation (i.e., PET from other research) which when combined with this study would be above the allowable limits.
11. Positive urine drug screen.
12. Pregnancy or breast feeding.
13. Inability to lie flat on camera bed for about 2.5 h

Healthy Subjects:

1. Any current Axis I diagnosis; and any past or present substance abuse other than a total lifetime use of cannabis of less than 10 times and no cannabis use within the last 3 months.
2. Family history of schizophrenia, schizophreniform disorder, or schizo-affective disorder.
3. Clinically significant laboratory abnormalities.
4. Recent heavy use of alcohol. That is, subjects must have an alcohol audit score of less than or equal to 9. In addition, subjects must agree not to consume any alcohol in the three days prior to the PET scan.
5. Psychotropic medication use (including benzodiazepines and illicit drugs) during the 28 days (42 day for fluoxetine) prior to the PET scan.
6. Serious medical problems.
7. Positive test for HIV.
8. Metallic foreign bodies that would be affected by the MRI magnet, or fear of enclosed spaces likely to make the subject unable to undergo an MRI scan.
9. Head trauma resulting in a period of unconsciousness lasting longer than 10 minutes.
10. History of fetal alcohol syndrome or other neurodevelopmental disorder.
11. History of seizures, other than in childhood and related to fever.
12. Recent exposure to radiation (i.e., PET from other research) which when combined with this study would be above the allowable limits.
13. Positive urine drug screen.
14. Pregnancy or breast feeding.
15. Inability to lie flat on camera bed for about 2.5 h

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2010-02-01; Study Completion 2012-09-20

PRIMARY OUTCOMES:
Brain distribution volume of 18F-FMPEP-d2.

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Abi-Dargham A, Rodenhiser J, Printz D, Zea-Ponce Y, Gil R, Kegeles LS, Weiss R, Cooper TB, Mann JJ, Van Heertum RL, Gorman JM, Laruelle M. Increased baseline occupancy of D2 receptors by dopamine in schizophrenia. Proc Natl Acad Sci U S A. 2000 Jul 5;97(14):8104-9. doi: 10.1073/pnas.97.14.8104. PMID 10884434
- [Background] Andreasson S, Allebeck P, Engstrom A, Rydberg U. Cannabis and schizophrenia. A longitudinal study of Swedish conscripts. Lancet. 1987 Dec 26;2(8574):1483-6. doi: 10.1016/s0140-6736(87)92620-1. PMID 2892048
- [Background] Arseneault L, Cannon M, Poulton R, Murray R, Caspi A, Moffitt TE. Cannabis use in adolescence and risk for adult psychosis: longitudinal prospective study. BMJ. 2002 Nov 23;325(7374):1212-3. doi: 10.1136/bmj.325.7374.1212. No abstract available. PMID 12446537